CLINICAL TRIAL: NCT06617897
Title: A Phase 3, Single-center, Randomized, Controlled Clinical Study to Investigate the Efficacy of Fibrinogen Concentrate (CSL511) in Subjects With Pseudomyxoma Peritonei Undergoing Cytoreductive Surgery
Brief Title: Phase 3 Study of Fibrinogen Concentrate (CSL511) in Subjects With Pseudomyxoma Peritonei Undergoing Cytoreductive Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSL511_3003
Record Dates: First submitted 2024-09-24; First posted 2024-10-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Acquired Fibrinogen Deficiency
Keywords: Fibrinogen deficiency; Pseudomyxoma peritonei; Cytoreductive surgery; Hyperthermic intraperitoneal chemotherapy; Blood coagulation disorder
MeSH Terms: conditions — Afibrinogenemia; Pseudomyxoma Peritonei; Blood Coagulation Disorders | interventions — cryoprecipitate coagulum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSL511 (Experimental)
  Interventions: Biological: CSL511 Fibrinogen concentrate (human)
- Cryoprecipitate (Active Comparator)
  Interventions: Biological: Cryoprecipitate

INTERVENTIONS:
Biological: CSL511 Fibrinogen concentrate (human) — CSL511 will be prepared in sterile water for injection and administered as an intravenous (IV) infusion.
  Arms: CSL511
Biological: Cryoprecipitate — Cryoprecipitate will be administered via IV infusion.
  Arms: Cryoprecipitate

SUMMARY:
This study is a phase 3, prospective, single center, randomized, open label, controlled, parallel arm, interventional study to investigate the efficacy and safety of CSL511, in participants undergoing cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC) for pseudomyxoma peritonei (PMP) with predicted intraoperative blood loss of greater than or equal to (>=) 2 liter (L). Eligible participants will be randomized in a 1:1 ratio to 1 of 2 treatment arms, to receive CSL511 or cryoprecipitate.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 18 years at the time of providing written informed consent.
* Diagnosis of PMP requiring CRS with HIPEC.
* Bleeding risk: Predicted intraoperative blood loss of >=2L, assessed within 60 and 100 mins after start of study surgery (assessment made before 2 L of blood is lost)

Exclusion Criteria:

* Confirmed or suspected congenital or acquired coagulation disorder or a prothrombotic disorder
* Myocardial infarction, acute coronary syndrome, or stroke within 2 months before study surgery.
* Known history of chronic hepatitis.
* Clopidogrel or ticagrelor administration within 5 days before study surgery.
* Prasugrel administration within 7 days before study surgery.
* Oral factor Xa inhibitor administration within 2 days before study surgery.
* Glycoprotein IIb / IIIa antagonist administration within 24 hours before study surgery.
* Oral direct thrombin inhibitor administration within 3 days before study surgery.
* Vitamin K antagonists within 5 days before study surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with overall hemostatic success | During surgery to 24 hours after surgery
  Overall hemostatic success will be assessed by an independent data monitoring and efficacy adjudication committee (IDMEAC). The IDMEAC will assess the overall efficacy based on a composite of intraoperative and postoperative hemostasis using a 4-point scale, where ratings correspond to excellent or good (hemostatic success) or moderate or none (hemostatic failure).

SECONDARY OUTCOMES:
Number of participants with treatment-emergent (TE): adverse events (AEs), serious AEs (SAEs), and AEs of special interest (AESIs) | Up to 30 days after IV infusion
  The TE AESIs include thromboembolic events, viral transmission/seroconversion, and anaphylaxis and severe hypersensitivity/severe allergic reactions.
Number of participants with intraoperative hemostatic efficacy | During surgery
  Intraoperative hemostatic efficacy will be assessed by the surgeon and anesthesiologist using an objective 4-point hemostatic efficacy scale, where ratings correspond to excellent or good (hemostatic success) or moderate or none (hemostatic failure).
Number of participants with postoperative hemostatic efficacy | Up to 24 hours after surgery
  Postoperative hemostatic efficacy will be assessed by a hematologist using an objective 4-point hemostatic efficacy scale, where ratings correspond to excellent or good (hemostatic success) or moderate or none (hemostatic failure).
Plasma fibrinogen concentration | During surgery, at the end of surgery and up to 24 hours after start of surgery
Mean total dose of fibrinogen administered | During surgery, at the end of surgery and up to 24 hours after start of surgery
Number of doses of fibrinogen administered | During surgery, at the end of surgery and up to 72 hours after start of surgery
Duration of surgery | During surgery
Intraoperative blood loss | During surgery
Intraoperative requirements for blood products | During surgery
  Blood products include fresh frozen plasma, red blood cells, and platelets.
Postoperative blood loss | Up to 48 hours after start of surgery
Postoperative requirements for blood products | Up to 9 days after surgery
  Blood products include fresh frozen plasma, red blood cells, and platelets.
Number of participants with reoperation (for bleeding) | Up to 30 days after surgery
Number of participants with reoperation (for reasons other than bleeding) | Up to 30 days after surgery
Duration of mechanical ventilation | Up to 30 days after surgery
Duration of intensive care unit (ICU) stay | Up to 30 days after surgery
Duration of hospital stay | Up to 30 days after surgery
21-day mortality | Up to 21 days after surgery
In-hospital mortality | Up to 30 days after surgery
Time between placing the investigational product (IP) order to administration | During surgery
  The following time to event parameters will be assessed: time between when IP is ordered and when IP is ready to administer in the operating room and time between when IP is ordered and start of IP administration.
Prothrombin time and activated partial thromboplastin time | Up to 8 days after surgery
Coagulation parameter profile | Up to 8 days after surgery
  The following coagulation parameter profiles will be assessed: thrombin generation marker, protein C and S, antithrombin and alpha 2-antiplasmin.
Coagulation factor profile | Up to 8 days after surgery
  The following coagulation factor profiles will be assessed: fibrinogen, factor VIII (FVIII):C, von Willebrand ristocetin cofactor (VWF:Rco) and factor XIII (FXIII).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — CSL Behring
Locations (1):
- Basingstoke and North Hampshire Hospital, Basingstoke, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
CSL will consider on a case-by-case basis requests to share Individual Patient Data (IPD) with external bona-fide, qualified scientific and medical researchers. For information on the process and requirements for submitting a voluntary data sharing request for IPD, please contact CSL at clinicaltrials@cslbehring.com.
Supporting Information: Study Protocol, SAP
Time Frame: Requests for IPD will generally be considered once review by major regulatory authorities (ie FDA, EMA) is complete and the primary publication is available
Access Criteria: Proposed research should seek to answer a previously unanswered important medical or scientific question.
  Applicable country specific privacy and other laws and regulations will be considered and may prevent sharing of IPD.
  If the request is approved and the researcher has executed an appropriate data sharing agreement, IPD that has been appropriately anonymized will be available.